CLINICAL TRIAL: NCT00832429
Title: Sentinel Lymph Node Localization and Biopsy for Sebaceous Gland Carcinoma of the Eyelid
Brief Title: Lymph Node Mapping in Finding Metastatic Disease in Patients With Sebaceous Gland Cancer of the Eyelid
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-0266; NCI-2011-01097 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2008-0266 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Eyelid Sebaceous Gland Carcinoma
MeSH Terms: interventions — Sentinel Lymph Node Biopsy; Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Diagnostic (SLN localization and biopsy) (Experimental): Patients receive technetium Tc 99m sulfur colloid ID and then undergo lymph node mapping and SLN biopsy.
  Interventions: Procedure: Lymph Node Mapping; Procedure: Sentinel Lymph Node Biopsy; Drug: Technetium Tc-99m Sulfur Colloid

INTERVENTIONS:
Procedure: Lymph Node Mapping — Undergo lymph node mapping
  Other Names: lymphatic mapping
Procedure: Sentinel Lymph Node Biopsy — Undergo SLN biopsy
  Other Names: Sentinel Node Biopsy; Sentinel node biopsy alone; SLNB; SNB
Drug: Technetium Tc-99m Sulfur Colloid — Given ID
  Other Names: Tc 99m Sulfur Colloid; Tc-99m SC; Technetium Tc 99m Sulfur Colloid

SUMMARY:
This phase II trial studies how well lymph node mapping works in finding disease that has spread from the place where it started to other places in the body in patients with sebaceous gland cancer of the eyelid. Lymph node mapping may help in planning surgery to remove cancer and affected lymph nodes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Identify the rate of SLN (sentinel lymph node) positivity for eyelid sebaceous gland carcinomas.

II. Identify the false negative events associated with SLN biopsy for sebaceous gland carcinomas.

SECONDARY OBJECTIVE:

I. Record any side effects associated with SLN biopsy for sebaceous gland carcinoma of the eyelid.

OUTLINE:

Patients receive technetium Tc 99m sulfur colloid intradermally (ID) and then undergo lymph node mapping and SLN biopsy.

After completion of study treatment, patients are followed up every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Possible or suspicious sebaceous gland carcinoma of the eyelid
* A CXR (chest x-ray), liver enzymes, and a head and neck computed tomography (CT), a single photon emission computed tomography (SPECT/CT) or magnetic resonance imaging (MRI) and an ultrasound negative for clinical evidence of metastasis
* Patient provided written informed consent; in the event that non-English speaking participants are eligible for this study, a short form (if applicable) or an informed consent document (ICD) in their language, will be utilized and completed in accordance with the M.D. Anderson Cancer Center (MDACC) Policy for Consenting Non-English Speaking Participants

Exclusion Criteria:

* Pregnant or nursing females

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02-25 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bita M Esmaeli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with sebaceous carcinoma of the eyelid treated at MDA from 2009-2021
Groups:
- Patients With Sebaceous Carcinoma Who Opted to Receive SLN Biopsy: There was only one arm to the study as this was a feasibility study
Period: Overall Study
Arm/Group | Patients With Sebaceous Carcinoma Who Opted to Receive SLN Biopsy
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Sentinel Lymph Node Localization and Biopsy for Sebaceous Gland Carcinoma of the Eyelid: Patients with sebaceous carcinoma who opted to receive SLN biopsy
Arm/Group | Sentinel Lymph Node Localization and Biopsy for Sebaceous Gland Carcinoma of the Eyelid
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Sentinel Lymph Node Positivity
Description: Number of patients who had a positive sentinel lymph node
Time Frame: One year after the surgical procedure under study.
Measure: Count of Participants; unit: Participants
Arm/Group | Sentinel Lymph Node Localization and Biopsy for Sebaceous Gland Carcinoma of the Eyelid
Number analyzed (Participants) | 20
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Sentinel Lymph Node Localization and Biopsy for Sebaceous Gland Carcinoma of the Eyelid
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-27): https://cdn.clinicaltrials.gov/large-docs/29/NCT00832429/Prot_SAP_000.pdf